CLINICAL TRIAL: NCT02965066
Title: Clinical Study Investigating Safety and Performance of a New Urinary Intermittent Catheter in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CP269
Record Dates: First submitted 2016-11-11; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Incontinence, Urinary
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Coloplast Test catheter; then Speedicath catheter (Experimental): The subjects allocated to this arm first test Coloplast Test catheter and after cross over test the comparator speedicath catheter
  Interventions: Device: Coloplast Test Catheter; Device: Coloplast Speedicath
- First Speedicath catheter; then Coloplast Test catheter (Experimental): The subjects allocated to this arm first test Speedicath catheter and after cross over test the Coloplast test catheter
  Interventions: Device: Coloplast Test Catheter; Device: Coloplast Speedicath

INTERVENTIONS:
Device: Coloplast Test Catheter — Newly developed intermittent catheter
Device: Coloplast Speedicath — Marketed Coloplast Speedicath catheter

SUMMARY:
The aim of the study is to test the performance and safety of a newly developed intermittent catheter in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and signed letter of authority
2. Be at least 18 years of age and have full legal capacity
3. Be a male
4. Willing to refrain from using analgetics up to 24 hours prior to catheterization visits
5. Have a negative urine multistix - erythrocytes (Microscopic haematuria)
6. Have a negative urine multistix:

   * Leukocytes
   * Nitrite Or if positive, subsequent negative for bacterial growth in urine culture

Exclusion Criteria:

1. Abnormalities, diseases or surgical procedures performed in the lower urinary tract
2. Symptoms of urinary tract infections (at least one of the following: frequent urination, stinging or pain at urination)
3. Participating in other clinical investigations related to urinary tracts system during this investigation (inclusion to termination) or have previously participated in this investigation
4. Known hypersensitivity toward any of the test products -

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Pain | 1 day
  The VAS scale is used to measure the pain experienced by the subjects at catheterisation

CONTACTS AND LOCATIONS:
Overall Officials: Per Bagi, MD, Principal Investigator — MD at the clinic of urology at Rigshospitalet
Locations (1):
- Rigshospitalet, Coppenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No